CLINICAL TRIAL: NCT03807453
Title: Comparison of Scalp Microbiota of the Patients With Psoriasis Vulgaris and Seborrheic Dermatitis
Brief Title: Comparison of Scalp Microbiota of the Psoriasis and Seborrheic Dermatitis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Turkish Dermatology Association (Unknown)
Responsible Party: Principal Investigator, Melek Aslan Kayıran, Dermatologist, M.D., Istanbul Medeniyet University
Other Study IDs: IstanbulMU2
Record Dates: First submitted 2019-01-05; First posted 2019-01-17 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis Vulgaris; Seborrheic Dermatitis; Microbial Colonization
Keywords: Psoriasis Vulgaris; Seborrheic Dermatitis; Scalp; Microbiome
MeSH Terms: conditions — Dermatitis, Seborrheic; Communicable Diseases | interventions — Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Psoriasis Vulgaris patients-Lesion
  Interventions: Other: Microbiota
- Psoriasis Vulgaris patients-Lesion free
  Interventions: Other: Microbiota
- Seborrheic Dermatitis-Lesion
  Interventions: Other: Microbiota
- Seborrheic Dermatitis-Lesion free
  Interventions: Other: Microbiota
- Control Group
  Interventions: Other: Microbiota

INTERVENTIONS:
Other: Microbiota — The scalp microbiota

SUMMARY:
A sterile swap specimen taken from the scalp of the patients with psoriasis vulgaris or seborrheic dermatitis and the volunteer control group will be examined in our study. The examples of the microbiota of the patients will be taken both the lesional scalp and the lesion-free part of the scalp. Then, the microbiota differences between the lesioned scalp and the lesion-free scalp of both groups, and the microbiome differences between the two groups and the control group will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with scalp psoriasis
2. Patients with seborrheic dermatitis
3. Agree to participate in research 4 - Do not use any drugs for their disease topically or systemically for two months

Exclusion Criteria:

1. Patients who do not want to participate in the study
2. Patients with psoriasis vulgaris or seborrheic dermatitis that does not effect scalp.
3. Those with chronic diseases that may affect skin microbiome
4. Patients using antibiotics, antifungal or antiviral therapy for any reason for the last one month.
5. Patients who are using topical or systemic drugs for their illness

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: primary care clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
The scalp microbiota of the patients with psoriasis and seborrheic dermatitis | 6 months
  The aim of this study is to compare the scalp microbiota of psoriasis vulgaris and seborrheic dermatitis both the lesion and lesion-free parts and also the control group and to assess their role on etiopathogenesis. Determining the microbiota of this region which is frequently involved and resistant to treatment may change the treatment approach. In addition, scalp microbiome of seborrheic dermatitis may be a causal factor of rapid relapse after treatment.
  The similarities between the microbiota of the psoriasis vulgaris and seborrheic dermatitis cases with only scalp involvement can guide us not only for the diagnosis but also the treatment. There are a few reports about the role of Malassezia subgroups in the pathogenesis, but it is known that there are many different flora members on the scalp. Exposing these can change both our diagnosis and treatment options.

SECONDARY OUTCOMES:
The differences between the scalp microbiota of different countries | 6 months
  Does the microbiota of the patients change between the countries? To our knowledge, there is no similar studies in present. Presenting the scalp microbiome of Turkish population can be a start to understand whether there is a difference in terms of the countries.

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Aslan Kayıran, Istanbul, Turkey (Türkiye)